CLINICAL TRIAL: NCT02846714
Title: FLARE: Family Lifestyle Actions and Risk Education Study for Children With a Familial Risk for Melanoma
Brief Title: Family Lifestyle Actions and Risk Education Study
Acronym: FLARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yelena Wu, Assistant Professor, Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00090292; K07CA196985 (NIH)
Record Dates: First submitted 2016-07-17; First posted 2016-07-27 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Melanoma; Child
Keywords: Education; Prevention and Control; Behavioral Research
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FLARE intervention (Experimental): All FLARE participants enrolled will receive the intervention
  Interventions: Behavioral: FLARE

INTERVENTIONS:
Behavioral: FLARE

SUMMARY:
The overall purpose of this study is to test the feasibility, acceptability, and preliminary efficacy of a family-focused behavioral intervention ("FLARE", which stands for Family Lifestyle Actions and Risk Education) that aims to improve adherence to melanoma preventive behaviors among children at elevated risk for the disease.

DETAILED DESCRIPTION:
Test the feasibility and acceptability of FLARE, a family-focused behavioral intervention that is designed to improve and maintain adherence to photoprotection (e.g., use of sunscreen) and screening (e.g., implementation of self skin exams). We expect that the feasibility of the intervention will be supported by at least 75% of participants attending at least 3 intervention sessions. We also expect that the acceptability of the intervention (e.g., overall satisfaction, ease of participation, perceived utility of intervention) will be supported by mean ratings that indicate adequate levels of acceptability across participants (e.g., mean rating of "satisfied" or "very satisfied" for overall satisfaction).

Pilot test the efficacy of the FLARE intervention with children at elevated risk for melanoma and their primary caregiver.

We will also explore the potential impact of the FLARE intervention on melanoma preventive behaviors among siblings of the child who receives the intervention, as well as the child's other parent/caregiver (if another parent/caregiver is available).

ELIGIBILITY:
Inclusion Criteria:

Children

* Are 8-17 years old AND
* Are at risk for melanoma due to having a first degree relative with a history of melanoma and/or at least 3 second or third degree relatives on the same side of the family with a history of melanoma AND/OR
* Have personally received genetic testing for the CDKN2A/p16 genetic mutation and/or has one or more family members who received CDKN2A/p16 testing

Adults

* Are at least 18 years old AND
* Are the primary caregiver for the child participating in the study (defined as the individual who is responsible for daily implementation of health-related tasks for the child) AND
* Have at least one child under age 18 who is living in the same household AND
* Have a personal history of melanoma and/or family history of melanoma) AND/OR
* Have personally received genetic testing for the CDKN2A/p16 genetic mutation and/or has one or more family members who received CDKN2A/p16 testing

Exclusion Criteria:

* Individuals who do not speak, read/write English will be excluded because FLARE involves regular interaction between study staff and research participants in English and completion of study questionnaires and interviews in English

Ages: 8 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-07; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yelena Wu, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glanz K, Yaroch AL, Dancel M, Saraiya M, Crane LA, Buller DB, Manne S, O'Riordan DL, Heckman CJ, Hay J, Robinson JK. Measures of sun exposure and sun protection practices for behavioral and epidemiologic research. Arch Dermatol. 2008 Feb;144(2):217-22. doi: 10.1001/archdermatol.2007.46. PMID 18283179
- [Background] Weinstock MA, Risica PM, Martin RA, Rakowski W, Smith KJ, Berwick M, Goldstein MG, Upegui D, Lasater T. Reliability of assessment and circumstances of performance of thorough skin self-examination for the early detection of melanoma in the Check-It-Out Project. Prev Med. 2004 Jun;38(6):761-5. doi: 10.1016/j.ypmed.2004.01.020. PMID 15193896
- [Background] Gwadry-Sridhar F, Guyatt GH, Arnold JM, Massel D, Brown J, Nadeau L, Lawrence S. Instruments to measure acceptability of information and acquisition of knowledge in patients with heart failure. Eur J Heart Fail. 2003 Dec;5(6):783-91. doi: 10.1016/s1388-9842(03)00158-2. PMID 14675857
- [Background] Kothe EJ, Mullan BA. Acceptability of a theory of planned behaviour email-based nutrition intervention. Health Promot Int. 2014 Mar;29(1):81-90. doi: 10.1093/heapro/das043. Epub 2012 Aug 31. PMID 22942273
- [Background] Gage H, Grainger L, Ting S, Williams P, Chorley C, Carey G, Borg N, Bryan K, Castleton B, Trend P, Kaye J, Jordan J, Wade D. Specialist rehabilitation for people with Parkinson's disease in the community: a randomised controlled trial. Southampton (UK): NIHR Journals Library; 2014 Dec. Available from http://www.ncbi.nlm.nih.gov/books/NBK263782/ PMID 25642574
- [Background] Stump, T. K., Aspinwall, L. G., Taber, J. M., Edwards, R., & Leachman, S. A. Validation of the Protection-Adjusted Length of Exposure (PALE) Index - A New Self-Report Measure of UVR Exposure (2014, April). Paper presented at the annual meeting of the Society of Behavioral Medicine, Philadelphia, PA.
- [Derived] Wu YP, Boucher K, Hu N, Hay J, Kohlmann W, Aspinwall LG, Bowen DJ, Parsons BG, Nagelhout ES, Grossman D, Mooney K, Leachman SA, Tercyak KP. A pilot study of a telehealth family-focused melanoma preventive intervention for children with a family history of melanoma. Psychooncology. 2020 Jan;29(1):148-155. doi: 10.1002/pon.5232. Epub 2019 Nov 10. PMID 31520429

RESULTS

PARTICIPANT FLOW:
Groups:
- FLARE Intervention: FLARE participants enrolled
Period: Overall Study
Arm/Group | FLARE Intervention
Started | 42
Completed | 36
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Parent participant age | 41.3 (5.0)
  Child participant age | 11.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 39
  Race/Ethnicity: White Hispanic | 2
  Race/Ethnicity: Biracial | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Retained Throughout Intervention as Assessed by Session Attendance Recorded by Interventionist
Description: Session attendance will be recorded by the interventionist at each scheduled session. The percent of participants who are retained throughout the 3 session intervention will be calculated.
Time Frame: Week 9 (post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Participants | 36

2. Secondary Outcome: Photoprotective Behaviors Assessed With the Sun Habits Survey
Description: "These next questions ask about what you have done in the past month if you were outdoors in the sun for 15 minutes or more. How often did you..." Minimum value = 1; Maximum value = 5; Higher scores indicate a better outcome
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: Outcomes for parents (n=21) are from parent self-report of behavior; outcomes for children (n=21) are from parent report on child's behavior
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
units on a scale
  Wk 1 - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 1 - Parent - use sunscreen | 4.29 (.56)
  Wk 1 - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 1 - Parent - reapply sunscreen | 3.56 (.86)
  Wk 1 - Parent - wear shirt w/ long sleeves: number analyzed (Participants) | 21
  Wk 1 - Parent - wear shirt w/ long sleeves | 2.29 (1.06)
  Wk 1 - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 1 - Parent - wear long pants or skirt | 2.76 (1.14)
  Wk 1 - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 1 - Parent - wear a wide-brimmed hat | 2.71 (1.19)
  Wk 1 - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 1 - Parent - stay in shade | 3.38 (.92)
  Wk 1 - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 1 - Parent - avoid sun 10am-4pm | 3.00 (.84)
  Wk 1 - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 1 - Parent - wear sunglasses | 4.10 (1.26)
  Wk 1 - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 1 - Parent - intentionally tan outdoors | 1.14 (.48)
  Wk 1 - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 1 - Parent - use an indoor tanning bed | 1.06 (.24)
  Wk 3 - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 3 - Parent - use sunscreen | 4.00 (1.14)
  Wk 3 - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 3 - Parent - reapply sunscreen | 2.93 (1.39)
  Wk 3 - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 3 - Parent - wear shirt w/long sleeves | 2.61 (.98)
  Wk 3 - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 3 - Parent - wear long pants or skirt | 3.22 (1.17)
  Wk 3 - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 3 - Parent - wear a wide-brimmed hat | 2.11 (.96)
  Wk 3 - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 3 - Parent - stay in shade | 3.44 (.92)
  Wk 3 - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 3 - Parent - avoid sun 10am-4pm | 2.83 (1.10)
  Wk 3 - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 3 - Parent - wear sunglasses | 4.00 (1.28)
  Wk 3 - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 3 - Parent - intentionally tan outdoors | 1.11 (.32)
  Wk 3 - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 3 - Parent - use an indoor tanning bed | 1.00 (0)
  Wk 5 - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 5 - Parent - use sunscreen | 3.68 (1.29)
  Wk 5 - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 5 - Parent - reapply sunscreen | 3.50 (1.03)
  Wk 5 - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 5 - Parent - wear shirt w/long sleeves | 2.21 (1.03)
  Wk 5 - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 5 - Parent - wear long pants or skirt | 3.00 (1.11)
  Wk 5 - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 5 - Parent - wear a wide-brimmed hat | 2.05 (1.08)
  Wk 5 - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 5 - Parent - stay in shade | 3.37 (.76)
  Wk 5 - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 5 - Parent - avoid sun 10am-4pm | 3.00 (1.20)
  Wk 5 - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 5 - Parent - wear sunglasses | 3.89 (1.33)
  Wk 5 - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 5 - Parent - intentionally tan outdoors | 1.05 (.23)
  Wk 5 - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 5 - Parent - use an indoor tanning bed | 1.00 (0)
  Wk 7 - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 7 - Parent - use sunscreen | 3.63 (1.46)
  Wk 7 - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 7 - Parent - reapply sunscreen | 3.00 (1.47)
  Wk 7 - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 7 - Parent - wear shirt w/long sleeves | 2.44 (1.32)
  Wk 7 - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 7 - Parent - wear long pants or skirt | 3.37 (1.36)
  Wk 7 - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 7 - Parent - wear a wide-brimmed hat | 2.19 (1.22)
  Wk 7 - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 7 - Parent - stay in shade | 3.44 (1.03)
  Wk 7 - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 7 - Parent - avoid sun 10am-4pm | 2.94 (1.34)
  Wk 7 - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 7 - Parent - wear sunglasses | 4.00 (1.41)
  Wk 7 - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 7 - Parent - intentionally tan outdoors | 1.00 (0)
  Wk 7 - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 7 - Parent - use an indoor tanning bed | 1.00 (0)
  Wk 9 - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 9 - Parent - use sunscreen | 3.67 (1.33)
  Wk 9 - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 9 - Parent - reapply sunscreen | 3.33 (1.40)
  Wk 9 - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 9 - Parent - wear shirt w/long sleeves | 2.72 (1.02)
  Wk 9 - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 9 - Parent - wear long pants or skirt | 3.40 (1.15)
  Wk 9 - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 9 - Parent - wear a wide-brimmed hat | 1.89 (.9)
  Wk 9 - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 9 - Parent - stay in shade | 3.33 (.84)
  Wk 9 - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 9 - Parent - avoid sun 10am-4pm | 3.33 (.97)
  Wk 9 - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 9 - Parent - wear sunglasses | 4.00 (1.33)
  Wk 9 - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 9 - Parent - intentionally tan outdoors | 1.06 (.24)
  Wk 9 - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 9 - Parent - use an indoor tanning bed | 1.00 (0)
  Wk 13 - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 13 - Parent - use sunscreen | 3.63 (1.46)
  Wk 13 - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 13 - Parent - reapply sunscreen | 3.15 (1.46)
  Wk 13 - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 13 - Parent - wear shirt w/long sleeves | 3.25 (1.18)
  Wk 13 - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 13 - Parent - wear long pants or skirt | 3.81 (1.17)
  Wk 13 - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 13 - Parent - wear a wide-brimmed hat | 1.94 (1.00)
  Wk 13 - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 13 - Parent - stay in shade | 3.44 (.96)
  Wk 13 - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 13 - Parent - avoid sun 10am-4pm | 2.94 (1.18)
  Wk 13 - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 13 - Parent - wear sunglasses | 3.94 (1.48)
  Wk 13 - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 13 - Parent - intentionally tan outdoors | 1.06 (.25)
  Wk 13 - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 13 - Parent - use an indoor tanning bed | 1.00 (0)
  Wk 1 - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 1 - Child - use sunscreen | 3.90 (.63)
  Wk 1 - Child - reapply sunscreen: number analyzed (Participants) | 21
  Wk 1 - Child - reapply sunscreen | 3.44 (1.04)
  Wk 1 - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 1 - Child - wear shirt w/long sleeves | 1.95 (.87)
  Wk 1 - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 1 - Child - wear long pants or skirt | 2.05 (1.02)
  Wk 1 - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 1 - Child - wear a wide-brimmed hat | 1.62 (.81)
  Wk 1 - Child - stay in shade: number analyzed (Participants) | 21
  Wk 1 - Child - stay in shade | 2.57 (1.17)
  Wk 1 - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 1 - Child - avoid sun 10am-4pm | 2.33 (1.11)
  Wk 1 - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 1 - Child - wear sunglasses | 1.81 (.75)
  Wk 1 - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 1 - Child - intentionally tan outdoors | 1.29 (.64)
  Wk 1 - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 1 - Child - use an indoor tanning bed | 1.00 (0)
  Wk 3 - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 3 - Child - use sunscreen | 3.88 (1.05)
  Wk 3 - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 3 - Child - wear shirt w/long sleeves | 2.11 (.68)
  Wk 3 - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 3 - Child - wear long pants or skirt | 2.22 (.81)
  Wk 3 - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 3 - Child - wear a wide-brimmed hat | 1.61 (.61)
  Wk 3 - Child - stay in shade: number analyzed (Participants) | 21
  Wk 3 - Child - stay in shade | 3.00 (1.03)
  Wk 3 - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 3 - Child - avoid sun 10am-4pm | 2.67 (1.24)
  Wk 3 - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 3 - Child - wear sunglasses | 1.89 (.96)
  Wk 3 - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 3 - Child - intentionally tan outdoors | 1.11 (.32)
  Wk 3 - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 3 - Child - use an indoor tanning bed | 1.00 (0)
  Wk 5 - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 5 - Child - use sunscreen | 4.11 (1.28)
  Wk 5 - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 5 - Child - wear shirt w/long sleeves | 2.05 (.97)
  Wk 5 - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 5 - Child - wear long pants or skirt | 2.32 (.89)
  Wk 5 - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 5 - Child - wear a wide-brimmed hat | 1.84 (1.30)
  Wk 5 - Child - stay in shade: number analyzed (Participants) | 21
  Wk 5 - Child - stay in shade | 3.21 (1.27)
  Wk 5 - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 5 - Child - avoid sun 10am-4pm | 2.95 (1.27)
  Wk 5 - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 5 - Child - wear sunglasses | 2.11 (1.37)
  Wk 5 - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 5 - Child - intentionally tan outdoors | 1.11 (.32)
  Wk 5 - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 5 - Child - use an indoor tanning bed | 1.00 (0)
  Wk 7 - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 7 - Child - use sunscreen | 4.07 (1.22)
  Wk 7 - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 7 - Child - wear shirt w/long sleeves | 2.44 (1.03)
  Wk 7 - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 7 - Child - wear long pants or skirt | 2.44 (.96)
  Wk 7 - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 7 - Child - wear a wide-brimmed hat | 1.75 (1.00)
  Wk 7 - Child - stay in shade: number analyzed (Participants) | 21
  Wk 7 - Child - stay in shade | 3.38 (1.67)
  Wk 7 - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 7 - Child - avoid sun 10am-4pm | 2.94 (1.69)
  Wk 7 - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 7 - Child - wear sunglasses | 1.75 (1.29)
  Wk 7 - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 7 - Child - intentionally tan outdoors | 1.00 (0)
  Wk 7 - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 7 - Child - use an indoor tanning bed | 1.00 (0)
  Wk 9 - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 9 - Child - use sunscreen | 3.94 (1.21)
  Wk 9 - Child - reapply sunscreen: number analyzed (Participants) | 21
  Wk 9 - Child - reapply sunscreen | 3.27 (1.39)
  Wk 9 - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 9 - Child - wear shirt w/long sleeves | 2.28 (.96)
  Wk 9 - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 9 - Child - wear long pants or skirt | 2.78 (1.26)
  Wk 9 - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 9 - Child - wear a wide-brimmed hat | 1.67 (1.24)
  Wk 9 - Child - stay in shade: number analyzed (Participants) | 21
  Wk 9 - Child - stay in shade | 3.44 (.98)
  Wk 9 - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 9 - Child - avoid sun 10am-4pm | 2.83 (1.04)
  Wk 9 - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 9 - Child - wear sunglasses | 1.67 (1.24)
  Wk 9 - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 9 - Child - intentionally tan outdoors | 1.00 (0)
  Wk 9 - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 9 - Child - use an indoor tanning bed | 1.00 (0)
  Wk 13 - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 13 - Child - use sunscreen | 3.69 (1.40)
  Wk 13 - Child - reapply sunscreen: number analyzed (Participants) | 21
  Wk 13 - Child - reapply sunscreen | 3.23 (1.54)
  Wk 13 - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 13 - Child - wear shirt w/long sleeves | 3.13 (.96)
  Wk 13 - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 13 - Child - wear long pants or skirt | 3.25 (1.07)
  Wk 13 - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 13 - Child - wear a wide-brimmed hat | 1.93 (1.03)
  Wk 13 - Child - stay in shade: number analyzed (Participants) | 21
  Wk 13 - Child - stay in shade | 3.06 (1.34)
  Wk 13 - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 13 - Child - avoid sun 10am-4pm | 2.75 (1.29)
  Wk 13 - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 13 - Child - wear sunglasses | 1.81 (1.28)
  Wk 13 - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 13 - Child - intentionally tan outdoors | 1.00 (0)
  Wk 13 - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 13 - Child - use an indoor tanning bed | 1.00 (0)

3. Secondary Outcome: Photoprotective Behaviors Assessed With the PALE Questionnaire
Description: Protection-Adjusted Length of Exposure Index (PALE) Assesses photoprotective behavior during reported activities to yield daily minutes of unprotected sun exposure during each time frame
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: Outcomes for parents (n=21) are from parent self-report of daily minutes of unprotected sun exposure; outcomes for children (n=21) are from parent report on child's daily minutes of unprotected sun exposure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
minutes
  Wk 1 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 1 - Parent - Weekday | 17.00 (29.46)
  Wk 1 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 1 - Parent - Weekend | 27.10 (36.73)
  Wk 3 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 3 - Parent - Weekday | 11.03 (15.23)
  Wk 3 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 3 - Parent - Weekend | 20.66 (43.53)
  Wk 5 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 5 - Parent - Weekday | 6.74 (10.83)
  Wk 5 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 5 - Parent - Weekend | 18.47 (31.02)
  Wk 7 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 7 - Parent - Weekday | 7.59 (24.29)
  Wk 7 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 7 - Parent - Weekend | 15.07 (33.00)
  Wk 9 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 9 - Parent - Weekday | .97 (2.49)
  Wk 9 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 9 - Parent - Weekend | 25.93 (40.28)
  Wk 13 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 13 - Parent - Weekday | 5.03 (16.17)
  Wk 13 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 13 - Parent - Weekend | 9.55 (14.22)
  Wk 1 - Child - Weekday: number analyzed (Participants) | 21
  Wk 1 - Child - Weekday | 37.43 (43.48)
  Wk 1 - Child - Weekend: number analyzed (Participants) | 21
  Wk 1 - Child - Weekend | 40.74 (45.50)
  Wk 3 - Child - Weekday: number analyzed (Participants) | 21
  Wk 3 - Child - Weekday | 12.79 (17.93)
  Wk 3 - Child - Weekend: number analyzed (Participants) | 21
  Wk 3 - Child - Weekend | 35.64 (55.01)
  Wk 5 - Child - Weekday: number analyzed (Participants) | 21
  Wk 5 - Child - Weekday | 18.63 (31.89)
  Wk 5 - Child - Weekend: number analyzed (Participants) | 21
  Wk 5 - Child - Weekend | 34.99 (56.88)
  Wk 7 - Child - Weekday: number analyzed (Participants) | 21
  Wk 7 - Child - Weekday | 26.87 (49.56)
  Wk 7 - Child - Weekend: number analyzed (Participants) | 21
  Wk 7 - Child - Weekend | 28.48 (44.26)
  Wk 9 - Child - Weekday: number analyzed (Participants) | 21
  Wk 9 - Child - Weekday | 24.23 (56.72)
  Wk 9 - Child - Weekend: number analyzed (Participants) | 21
  Wk 9 - Child - Weekend | 23.03 (53.07)
  Wk 13 - Child - Weekday: number analyzed (Participants) | 21
  Wk 13 - Child - Weekday | 32.93 (61.90)
  Wk 13 - Child - Weekend: number analyzed (Participants) | 21
  Wk 13 - Child - Weekend | 21.81 (42.29)

4. Secondary Outcome: Skin Self-exam Occurrence Assessed Via Questionnaire
Description: Number of participants who received a skin self-exam during each time frame
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: Outcomes for parents (n=21) are from parent self-report of skin self-exam; outcomes for children (n=21) are from parent report on child's skin self-exam
Measure: Count of Participants; unit: Participants
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Participants
  Wk 1 - Parent: number analyzed (Participants) | 21
  Wk 1 - Parent | 8
  Wk 3 - Parent: number analyzed (Participants) | 21
  Wk 3 - Parent | 6
  Wk 5 - Parent: number analyzed (Participants) | 21
  Wk 5 - Parent | 2
  Wk 7 - Parent: number analyzed (Participants) | 21
  Wk 7 - Parent | 4
  Wk 9 - Parent: number analyzed (Participants) | 21
  Wk 9 - Parent | 8
  Wk 13 - Parent: number analyzed (Participants) | 21
  Wk 13 - Parent | 8
  Wk 1 - Child: number analyzed (Participants) | 21
  Wk 1 - Child | 14
  Wk 3 - Child: number analyzed (Participants) | 21
  Wk 3 - Child | 13
  Wk 5 - Child: number analyzed (Participants) | 21
  Wk 5 - Child | 14
  Wk 7 - Child: number analyzed (Participants) | 21
  Wk 7 - Child | 12
  Wk 9 - Child: number analyzed (Participants) | 21
  Wk 9 - Child | 14
  Wk 13 - Child: number analyzed (Participants) | 21
  Wk 13 - Child | 13

5. Secondary Outcome: Skin Self-exam Occurrence Assessed Via Diary
Description: Number of participants who received a skin self-exam during each time frame interval
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: Outcomes for parents (n=21) are from parent self-report of skin self-exam; outcomes for children (n=21) are from child self-report of skin self-exam
Measure: Count of Participants; unit: Participants
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Participants
  Wk 1-3 - Parent: number analyzed (Participants) | 21
  Wk 1-3 - Parent | 6
  Wk 3-5 - Parent: number analyzed (Participants) | 21
  Wk 3-5 - Parent | 3
  Wk 5-7 - Parent: number analyzed (Participants) | 21
  Wk 5-7 - Parent | 3
  Wk 7-9 - Parent: number analyzed (Participants) | 21
  Wk 7-9 - Parent | 4
  Wk 9-13 - Parent: number analyzed (Participants) | 21
  Wk 9-13 - Parent | 5
  Wk 1-3 - Child: number analyzed (Participants) | 21
  Wk 1-3 - Child | 7
  Wk 3-5 - Child: number analyzed (Participants) | 21
  Wk 3-5 - Child | 4
  Wk 5-7 - Child: number analyzed (Participants) | 21
  Wk 5-7 - Child | 4
  Wk 7-9 - Child: number analyzed (Participants) | 21
  Wk 7-9 - Child | 4
  Wk 9-13 - Child: number analyzed (Participants) | 21
  Wk 9-13 - Child | 5

6. Secondary Outcome: Sunburn Occurrence Assessed Via Diary
Description: Number of participants who got a sunburn during each time frame interval
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: Outcomes for parents (n=21) are from parent self-report of sunburn occurrence; outcomes for children (n=21) are from child self-report of sunburn occurrence
Measure: Count of Participants; unit: Participants
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Participants
  Wk 1-3 - Parent: number analyzed (Participants) | 21
  Wk 1-3 - Parent | 0
  Wk 3-5 - Parent: number analyzed (Participants) | 21
  Wk 3-5 - Parent | 4
  Wk 5-7 - Parent: number analyzed (Participants) | 21
  Wk 5-7 - Parent | 2
  Wk 7-9 - Parent: number analyzed (Participants) | 21
  Wk 7-9 - Parent | 1
  Wk 9-13 - Parent: number analyzed (Participants) | 21
  Wk 9-13 - Parent | 2
  Wk 1-3 - Child: number analyzed (Participants) | 21
  Wk 1-3 - Child | 4
  Wk 3-5 - Child: number analyzed (Participants) | 21
  Wk 3-5 - Child | 2
  Wk 5-7 - Child: number analyzed (Participants) | 21
  Wk 5-7 - Child | 1
  Wk 7-9 - Child: number analyzed (Participants) | 21
  Wk 7-9 - Child | 2
  Wk 9-13 - Child: number analyzed (Participants) | 21
  Wk 9-13 - Child | 1

7. Secondary Outcome: Sunburn Occurrence Assessed Via Questionnaire
Description: Number of participants who received a sunburn during each time frame.
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: Outcomes for parents (n=21) are from parent self-report of sunburns; outcomes for children (n=21) are from parent report on child's sunburns
Measure: Count of Participants; unit: Participants
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Participants
  Wk 1 - Parent: number analyzed (Participants) | 21
  Wk 1 - Parent | 7
  Wk 3 - Parent: number analyzed (Participants) | 21
  Wk 3 - Parent | 0
  Wk 5 - Parent: number analyzed (Participants) | 21
  Wk 5 - Parent | 5
  Wk 7 - Parent: number analyzed (Participants) | 21
  Wk 7 - Parent | 2
  Wk 9 - Parent: number analyzed (Participants) | 21
  Wk 9 - Parent | 1
  Wk 13 - Parent: number analyzed (Participants) | 21
  Wk 13 - Parent | 1
  Wk 1 - Child: number analyzed (Participants) | 21
  Wk 1 - Child | 6
  Wk 3 - Child: number analyzed (Participants) | 21
  Wk 3 - Child | 2
  Wk 5 - Child: number analyzed (Participants) | 21
  Wk 5 - Child | 2
  Wk 7 - Child: number analyzed (Participants) | 21
  Wk 7 - Child | 1
  Wk 9 - Child: number analyzed (Participants) | 21
  Wk 9 - Child | 3
  Wk 13 - Child: number analyzed (Participants) | 21
  Wk 13 - Child | 1

8. Secondary Outcome: Ultraviolet Radiation (UVR) Exposure Assessed Via Dosimeter Device
Description: Change of weekly average UV intake from Week 1 (baseline) to Week 9 (post-intervention) and from Week 9 to Week 13 (1-month follow up)
Time Frame: Weeks 1 (baseline),9,13
Measure: Mean (Standard Error); unit: Joules/meter^2
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Joules/meter^2
  Wk 1 to Wk 9 | -1.38 (.33)
  Wk 9 to Wk 13 | .110 (.43)

9. Secondary Outcome: Ultraviolet Radiation (UVR) Exposure Assessed Via PALE Questionnaire
Description: Protection-Adjusted Length of Exposure Index (PALE) Assesses UVR exposure during reported activities to yield daily minutes of unprotected sun exposure during each time frame
Time Frame: Weeks 1 (baseline), 3,5,7,9,13
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
minutes
  Wk 1 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 1 - Parent - Weekday | 17.00 (29.46)
  Wk 1 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 1 - Parent - Weekend | 27.10 (36.73)
  Wk 3 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 3 - Parent - Weekday | 11.03 (15.23)
  Wk 3 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 3 - Parent - Weekend | 20.66 (43.53)
  Wk 5 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 5 - Parent - Weekday | 6.74 (10.83)
  Wk 5 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 5 - Parent - Weekend | 18.47 (31.02)
  Wk 7 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 7 - Parent - Weekday | 7.59 (24.29)
  Wk 7 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 7 - Parent - Weekend | 15.07 (33.00)
  Wk 9 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 9 - Parent - Weekday | .97 (2.49)
  Wk 9 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 9 - Parent - Weekend | 25.93 (40.28)
  Wk 13 - Parent - Weekday: number analyzed (Participants) | 21
  Wk 13 - Parent - Weekday | 5.03 (16.17)
  Wk 13 - Parent - Weekend: number analyzed (Participants) | 21
  Wk 13 - Parent - Weekend | 9.55 (14.22)
  Wk 1 - Child - Weekday: number analyzed (Participants) | 21
  Wk 1 - Child - Weekday | 37.43 (43.48)
  Wk 1 - Child - Weekend: number analyzed (Participants) | 21
  Wk 1 - Child - Weekend | 40.74 (45.50)
  Wk 3 - Child - Weekday: number analyzed (Participants) | 21
  Wk 3 - Child - Weekday | 12.79 (17.93)
  Wk 3 - Child - Weekend: number analyzed (Participants) | 21
  Wk 3 - Child - Weekend | 35.64 (55.01)
  Wk 5 - Child - Weekday: number analyzed (Participants) | 21
  Wk 5 - Child - Weekday | 18.63 (31.89)
  Wk 5 - Child - Weekend: number analyzed (Participants) | 21
  Wk 5 - Child - Weekend | 34.99 (56.88)
  Wk 7 - Child - Weekday: number analyzed (Participants) | 21
  Wk 7 - Child - Weekday | 26.87 (49.56)
  Wk 7 - Child - Weekend: number analyzed (Participants) | 21
  Wk 7 - Child - Weekend | 28.48 (44.26)
  Wk 9 - Child - Weekday: number analyzed (Participants) | 21
  Wk 9 - Child - Weekday | 24.23 (56.72)
  Wk 9 - Child - Weekend: number analyzed (Participants) | 21
  Wk 9 - Child - Weekend | 23.03 (53.07)
  Wk 13 - Child - Weekday: number analyzed (Participants) | 21
  Wk 13 - Child - Weekday | 32.93 (61.90)
  Wk 13 - Child - Weekend: number analyzed (Participants) | 21
  Wk 13 - Child - Weekend | 21.81 (42.29)

10. Secondary Outcome: Degree of Tan on Skin Assessed Via Reflectance Spectroscopy
Description: Mean degree of tan on skin assessed via reflectance spectroscopy of 4 different body parts (exposed wrist, outer arm, chin, and face) at each time frame. Measurements were taken using a spectrophotometer to quantify skin color. Melanin index values were recorded, with a higher value representing more melanin in the skin (i.e., darker skin).
Time Frame: Weeks 1 (baseline),9,13
Population: Outcomes for parents (n=21) are from parent's reflectance spectroscopy of skin; outcomes for children (n=21) are from child's reflectance spectroscopy of skin
Measure: Mean (Standard Deviation); unit: Melanin Index Values
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
Melanin Index Values
  Wk 1 - Parent - exposed wrist: number analyzed (Participants) | 21
  Wk 1 - Parent - exposed wrist | .59 (.33)
  Wk 1 - Parent - outer arm: number analyzed (Participants) | 21
  Wk 1 - Parent - outer arm | .49 (.22)
  Wk 1 - Parent - chin: number analyzed (Participants) | 21
  Wk 1 - Parent - chin | .77 (.21)
  Wk 1 - Parent - face: number analyzed (Participants) | 21
  Wk 1 - Parent - face | .71 (.23)
  Wk 9 - Parent - exposed wrist: number analyzed (Participants) | 21
  Wk 9 - Parent - exposed wrist | .57 (.21)
  Wk 9 - Parent - outer arm: number analyzed (Participants) | 21
  Wk 9 - Parent - outer arm | .56 (.21)
  Wk 9 - Parent - chin: number analyzed (Participants) | 21
  Wk 9 - Parent - chin | .73 (.17)
  Wk 9 - Parent - face: number analyzed (Participants) | 21
  Wk 9 - Parent - face | .69 (.18)
  Wk 13 - Parent - exposed wrist: number analyzed (Participants) | 21
  Wk 13 - Parent - exposed wrist | .56 (.20)
  Wk 13 - Parent - outer arm: number analyzed (Participants) | 21
  Wk 13 - Parent - outer arm | .55 (.18)
  Wk 13 - Parent - chin: number analyzed (Participants) | 21
  Wk 13 - Parent - chin | .73 (.16)
  Wk 13 - Parent - face: number analyzed (Participants) | 21
  Wk 13 - Parent - face | .70 (.20)
  Wk 1 - Child - exposed wrist: number analyzed (Participants) | 21
  Wk 1 - Child - exposed wrist | .44 (.25)
  Wk 1 - Child - outer arm: number analyzed (Participants) | 21
  Wk 1 - Child - outer arm | .36 (.36)
  Wk 1 - Child - chin: number analyzed (Participants) | 21
  Wk 1 - Child - chin | .39 (.33)
  Wk 1 - Child - face: number analyzed (Participants) | 21
  Wk 1 - Child - face | .43 (.29)
  Wk 9 - Child - exposed wrist: number analyzed (Participants) | 21
  Wk 9 - Child - exposed wrist | .44 (.32)
  Wk 9 - Child - outer arm: number analyzed (Participants) | 21
  Wk 9 - Child - outer arm | .32 (.32)
  Wk 9 - Child - chin: number analyzed (Participants) | 21
  Wk 9 - Child - chin | .31 (.34)
  Wk 9 - Child - face: number analyzed (Participants) | 21
  Wk 9 - Child - face | .39 (.34)
  Wk 13 - Child - exposed wrist: number analyzed (Participants) | 21
  Wk 13 - Child - exposed wrist | .38 (.26)
  Wk 13 - Child - outer arm: number analyzed (Participants) | 21
  Wk 13 - Child - outer arm | .28 (.36)
  Wk 13 - Child - chin: number analyzed (Participants) | 21
  Wk 13 - Child - chin | .25 (.26)
  Wk 13 - Child - face: number analyzed (Participants) | 21
  Wk 13 - Child - face | .34 (.27)

11. Secondary Outcome: Photoprotection Behavior Changes Assessed Via Questionnaire
Description: Mean difference for each photoprotection behavior from Week 1 (pre-intervention) to Week 9 (post-intervention) and from Week 9 to Week 13 (1 month follow-up).
  "These next questions ask about what you have done in the past month if you were outdoors in the sun for 15 minutes or more. How often did you..." Minimum value = 1; Maximum value = 5; A higher mean difference indicates a better outcome
Time Frame: Weeks 1,9,13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
score on a scale
  Wk 1-9 change - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - use sunscreen | -.61 (1.33)
  Wk 9-13 change - Parent - use sunscreen: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - use sunscreen | .06 (1.44)
  Wk 1-9 change - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - reapply sunscreen | -.27 (1.16)
  Wk 9-13 change - Parent - reapply sunscreen: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - reapply sunscreen | -.08 (1.26)
  Wk 1-9 change - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - wear shirt w/long sleeves | .50 (1.20)
  Wk9-13 change - Parent - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk9-13 change - Parent - wear shirt w/long sleeves | .56 (.73)
  Wk 1-9 change - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - wear long pants or skirt | .61 (1.04)
  Wk 9-13 change - Parent - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - wear long pants or skirt | .44 (.81)
  Wk 1-9 change - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - wear a wide-brimmed hat | -.72 (.83)
  Wk 9-13 change - Parent - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - wear a wide-brimmed hat | .06 (.57)
  Wk 1-9 change - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - stay in shade | -.11 (.68)
  Wk 9-13 change - Parent - stay in shade: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - stay in shade | .19 (.66)
  Wk 1-9 change - Parent - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - avoid sun 10am-4pm | .33 (.91)
  Wk 9-13 change - Parent - avoid sun 10am - 4pm: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - avoid sun 10am - 4pm | -.31 (.79)
  Wk 1-9 change - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - wear sunglasses | -.11 (.68)
  Wk 9-13 change - Parent - wear sunglasses: number analyzed (Participants) | 21
  Wk 9-13 change - Parent - wear sunglasses | .06 (.68)
  Wk1-9 change - Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk1-9 change - Parent - intentionally tan outdoors | -.11 (.32)
  Wk9-13 change- Parent - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk9-13 change- Parent - intentionally tan outdoors | 0 (0)
  Wk 1-9 change - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 1-9 change - Parent - use an indoor tanning bed | -.07 (.26)
  Wk9-13 change - Parent - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk9-13 change - Parent - use an indoor tanning bed | 0 (0)
  Wk 1-9 change - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 1-9 change - Child - use sunscreen | 0 (1.14)
  Wk 9-13 change - Child - use sunscreen: number analyzed (Participants) | 21
  Wk 9-13 change - Child - use sunscreen | -.33 (1.35)
  Wk 1-9 change - Child - reapply sunscreen: number analyzed (Participants) | 21
  Wk 1-9 change - Child - reapply sunscreen | -.20 (1.15)
  Wk 9-13 change - Child - reapply sunscreen: number analyzed (Participants) | 21
  Wk 9-13 change - Child - reapply sunscreen | .08 (1.19)
  Wk 1-9 change - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 1-9 change - Child - wear shirt w/long sleeves | .33 (1.24)
  Wk 9-13 change - Child - wear shirt w/long sleeves: number analyzed (Participants) | 21
  Wk 9-13 change - Child - wear shirt w/long sleeves | .94 (.93)
  Wk 1-9 change - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 1-9 change - Child - wear long pants or skirt | .72 (1.60)
  Wk 9-13 change - Child - wear long pants or skirt: number analyzed (Participants) | 21
  Wk 9-13 change - Child - wear long pants or skirt | .38 (1.09)
  Wk 1-9 change - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 1-9 change - Child - wear a wide-brimmed hat | 0 (.49)
  Wk 9-13 change - Child - wear a wide-brimmed hat: number analyzed (Participants) | 21
  Wk 9-13 change - Child - wear a wide-brimmed hat | .27 (.88)
  Wk 1-9 change - Child - stay in shade: number analyzed (Participants) | 21
  Wk 1-9 change - Child - stay in shade | .47 (1.07)
  Wk 9-13 change - Child - stay in shade: number analyzed (Participants) | 21
  Wk 9-13 change - Child - stay in shade | -.13 (1.19)
  Wk 1-9 change - Child - avoid sun 10am-4pm: number analyzed (Participants) | 21
  Wk 1-9 change - Child - avoid sun 10am-4pm | .28 (1.13)
  Wk 9-13 change - Child - avoid sun 10am - 4pm: number analyzed (Participants) | 21
  Wk 9-13 change - Child - avoid sun 10am - 4pm | .06 (.93)
  Wk 1-9 change - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 1-9 change - Child - wear sunglasses | -.41 (.80)
  Wk 9-13 change - Child - wear sunglasses: number analyzed (Participants) | 21
  Wk 9-13 change - Child - wear sunglasses | .40 (1.12)
  Wk 1-9 change - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk 1-9 change - Child - intentionally tan outdoors | -.22 (.55)
  Wk9-13 change - Child - intentionally tan outdoors: number analyzed (Participants) | 21
  Wk9-13 change - Child - intentionally tan outdoors | 0 (0)
  Wk 1-9 change - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 1-9 change - Child - use an indoor tanning bed | 0 (0)
  Wk 9-13 change - Child - use an indoor tanning bed: number analyzed (Participants) | 21
  Wk 9-13 change - Child - use an indoor tanning bed | 0 (0)

12. Secondary Outcome: Skin Self-exam Behavior Changes
Description: Mean difference for frequency of skin self-exam and thoroughness of skin self-exam (measured by number of body parts examined) from Week 1 (pre-intervention) to Week 9 (post-intervention) and from Week 9 to Week 13 (1 month follow-up). (SSE = skin self-exam)
  Change in frequency of SSE: "In the past month, how often did you check your skin for any new or changed moles or growths?" 1 = SSE less than once a month, 2 = SSE once a month, 3 = SSE more than once a month; higher mean difference indicates a better outcome.
  Change in thoroughness of SSE: "In the past month, which of the body parts listed below were checked for any new or changed moles or growths" Minimum value = 0 (checked 0 body parts during SSE); Maximum value = 15 (checked 15 body parts during SSE); higher mean difference indicates a better outcome
Time Frame: Weeks 1,9,13
Population: Outcomes for parents (n=21) are from parent self-report skin self-exam behavior changes; outcomes for children (n=21) are from parent report on child's skin self-exam behavior changes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
units on a scale
  Wk 1 to 9 change - Parent - frequency of SSE: number analyzed (Participants) | 21
  Wk 1 to 9 change - Parent - frequency of SSE | .25 (.50)
  Wk 9 to 13 change - Parent - frequency of SSE: number analyzed (Participants) | 21
  Wk 9 to 13 change - Parent - frequency of SSE | 0 (0)
  Wk 1 to 9 change - Parent - thoroughness of SSE: number analyzed (Participants) | 21
  Wk 1 to 9 change - Parent - thoroughness of SSE | 3.65 (9.09)
  Wk 9 to 13 change - Parent - thoroughness of SSE: number analyzed (Participants) | 21
  Wk 9 to 13 change - Parent - thoroughness of SSE | -1.06 (8.28)
  Wk 1 to 9 change - Child - frequency of SSE: number analyzed (Participants) | 21
  Wk 1 to 9 change - Child - frequency of SSE | -.31 (.87)
  Wk 9 to 13 change - Child - frequency of SSE: number analyzed (Participants) | 21
  Wk 9 to 13 change - Child - frequency of SSE | .27 (.46)
  Wk 1 to 9 change - Child - thoroughness of SSE: number analyzed (Participants) | 21
  Wk 1 to 9 change - Child - thoroughness of SSE | 3.83 (7.73)
  Wk 9 to 13 change - Child - thoroughness of SSE: number analyzed (Participants) | 21
  Wk 9 to 13 change - Child - thoroughness of SSE | -2.88 (7.75)

13. Secondary Outcome: Acceptability of Intervention Assessed Via Questionnaire
Description: "In these next 15 questions, we want to learn more about your thoughts about what you learned through the FLARE sessions you've had with us in-person and via WebEx or phone. Please indicate how much you agree with each statement." 15 total constructs summed, each was on the same 5 point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree).
  Minimum value = 1; Maximum Value = 75; higher score means a better outcome (better acceptability)
Time Frame: Week 9
Population: Outcomes for parents (n=21) are from parent self-report of acceptability; outcomes for children (n=21) are from child self-report of acceptability
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FLARE Intervention
Number analyzed (Participants) | 42
units on a scale
  Parent: number analyzed (Participants) | 21
  Parent | 51.67 (3.25)
  Child: number analyzed (Participants) | 21
  Child | 49.36 (5.31)

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | FLARE Intervention
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT02846714/Prot_SAP_000.pdf